CLINICAL TRIAL: NCT05397665
Title: A RandomIzed, Double-Blind, Placebo-CoNtrolled, Two-Part Study to Evaluate the Pharmacodynamic EffIcacy and Clinical Benefit of AT 007 in Patients With SoRbitol Dehydrogenase (SORD) DEficiency
Brief Title: Pharmacodynamic EffIcacy and Clinical Benefit of AT 007 in Patients With Sorbitol Dehydrogenase (SORD) Deficiency
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Applied Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-007-1005
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Neuropathy Caused by SORD Deficiency

STUDY DESIGN:
Intervention Model Description: Randomized, double blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: AT-007 and its matching placebo will have the same presentation, the same aspect and taste in order to be indistinguishable, and they will be supplied and used in the same conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AT-007 (Active Comparator): AT-007 is an Aldose reductase inhibitor
  Interventions: Drug: AT-007
- Placebo (Sham Comparator): Is an non-active control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AT-007 — AT-007, aldose reductase inhibitor
  Other Names: Govorestat
  Arms: AT-007
Drug: Placebo — Liquid oral suspension
  Other Names: Liquid oral vehicle suspension
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy and safety of AT-007 treatment in patients with SORD Deficiency. This randomized, double-blind study will assess the effect of AT-007 compared to Placebo in SORD Deficiency in patients for up to 24 months.

DETAILED DESCRIPTION:
This international, multi-center, randomized, double-blinded, placebo-controlled, phase 2-3 study is designed to assess the pharmacodynamic (PD) efficacy of AT-007 treatment, as well as the clinical benefit of long term administration to patients with SORD Deficiency utilizing a series of functional, patient-reported, and clinical outcomes measures.Safety and pharmacokinetics (PK) of AT-007 will also be evaluated. The study consists of Biomarker and Efficacy Assessments and an open-label extension (OLE) of active treatment for qualified patients.

Patients (18-55 years old) with SORD deficiency will be stratified according to their 10MWRT score (a single component of the CMT-FOM) and sex (male vs female). They will then be randomized in a 2:1 ratio to AT-007 20 mg/kg once daily (QD) or placebo.

The study will be conducted at up to 13 sites worldwide. A total of up to 72 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
2. Male and non-pregnant, non-lactating female patients between the ages of 18 and 55 years, inclusive.
3. Females must be of non-childbearing potential (defined as surgically sterile [i.e., had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy ≥6 months prior to the first dose of study drug] or postmenopausal for ≥1 year [confirmatory follicle stimulating hormone or FSH test results required] prior to the first dose of study drug) or agree to use an acceptable form of birth control from Screening until 30 days after the last dose of study drug.
4. Males must be unable to procreate (defined as surgically sterile [i.e., had a vasectomy ≥6 months prior to Screening]) or must agree to use an acceptable form of birth control from Screening through 30 days after the last dose of study drug.
5. Clinical diagnosis of CMT2 or dHMN due to SORD Deficiency confirmed by medical record or written communication by health care professional, elevated sorbitol level (>10,000 ng/mL), and gene analysis report indicating a biallelic mutation in SORD.
6. Patient may be on concomitant medications and dietary supplements; however, they must be on stable doses for at least 1 month prior to Screening and throughout the study. In addition, all over-the-counter (OTC) and/or prescription medications must be reviewed and approved by the Investigator.
7. Willing and able to be confined to the clinical research unit (CRU) as required by the protocol.

Exclusion Criteria:

1. 10MWRT classified as very severe disease (e.g. 10MWRT >15 seconds to complete OR unable to complete 10MWRT without the use of an assistive device such as a cane/walker/wheelchair).
2. History or presence of clinically significant hematopoietic, renal, hepatic, endocrine (e.g. diabetes), metabolic, pulmonary, neurological (e.g. other neuropathy, myopathy or neuromuscular disorder), psychiatric, cardiovascular, immunological, dermatological, or gastrointestinal diseases that are -at priori- altering the proper evaluation of the safety and efficacy of AT-007; conditions capable of altering the absorption, metabolism, or elimination of drugs; or conditions that constitute a risk factor when taking the study drug and/or impact the conduct or results of the study.
3. Body Mass Index (BMI) >35 kg/m2.
4. Clinically relevant underweight, weight loss suggestive of a pathology unrelated to SORD deficiency, or BMI < 17.5 kg/m2.
5. Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at Screening or previous treatment for hepatitis B, hepatitis C, or HIV infection.
6. Individuals who smoke or use tobacco or nicotine-containing products.
7. Pregnant, lactating, or not using/not willing to use appropriate means of contraception.
8. Any prior history of substance abuse (including alcohol) or treatment for such.
9. Positive urine drug screen (UDS) for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates) or cotinine.
10. Non-ambulatory disability.
11. Prior bilateral ankle stabilization surgery.
12. Impaired renal function or estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m2. Note: The eGFR is an estimation of renal function, and the ultimate decision of whether a patient has normal renal function (and can be included in the study) is at the discretion of the Investigator, assuming there are no safety concerns. Also, because eGFR can vary from day to day based on outside factors, patients can be re-screened for eGFR multiple times to understand the renal function of the patient.
13. Hemoglobin (Hgb) < 10.0 g/dL at Screening.
14. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin (except in case of Gilbert's syndrome) > 1.5 x upper limit of normal (ULN) at Screening.
15. Urinary albumin-to-creatinine ratio (UACR) > 30 mg/g at Screening in the presence of elevated creatinine (>2X ULN).
16. History or presence of cardiovascular disorders including myocardial infarction, stroke, uncontrolled hypertension (sitting blood pressure ≥140/90 mmHg), left ventricular (LV) hypertrophy, atrial fibrillation, or valvular heart disease considered clinically significant by the Principal Investigator (PI) and/or Sponsor medical representative.
17. Abnormal findings on the Screening 12-lead ECG, such as ST/T wave changes, pathological Q wave changes, or any rhythm other than normal sinus rhythm considered clinically significant by the PI and/or Sponsor medical representative.
18. Evidence of significant active hematological disease and/or cumulative blood donation of 1 unit (500 mL) or more including blood drawn during clinical studies in the last 3 months.
19. History of significant drug allergy or drug hypersensitivity.
20. Investigators, site personnel directly affiliated with this study, and their immediate families (defined as a spouse, parent, child, or sibling, whether biological or legally adopted).
21. Any other condition that, in the opinion of the Investigator, precludes the patient from following and completing the protocol.
22. A clinically significant abnormal finding on the physical exam/visual health assessment, medical history, ECG, or clinical laboratory results at Screening.
23. A significantly abnormal diet (per Investigator judgment) during the 4 weeks preceding the first dose of study drug.
24. Participation in another clinical study of a different investigational product within 30 days prior to the first dose of study drug.
25. Use of any OTC medication (including nutritional or dietary supplements, herbal preparations, or vitamins) ≤7 days prior to the first dose of study drug until the last dose of study drug without evaluation and approval by the Investigator.
26. Use of any prescription medication, except those allowed per protocol, from 30 days prior to the first dose of study drug until the last dose of study drug without evaluation and approval by the Investigator.
27. Treatment with any sensitive substrates of Breast Cancer Resistance Protein (BCRP) or potent inhibitors of BCRP.
28. Treatment with any sensitive substrates of cytochrome P450 3A4 (CYP3A4), CYP2B6, CYP2C19, or CYP1A2.
29. Treatment with any sensitive substrates of Organic Anion Transporter (OAT)1 and OAT3. Treatment with any drugs potentially associated with transaminase elevations. Potentially nephrotoxic drugs are prohibited.
30. Consumption of beverages or foods that contain alcohol, high levels of sorbitol, grapefruit, poppy seeds, broccoli, brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to the first dose of study drug through the last dose of study drug. Patients will be instructed not to consume any of the above products; however, allowance for sporadic consumption may be evaluated and approved by the Investigator based on the potential for interaction with the study drug. Not more than half cup of coffee per day should be consumed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
10-meter walk-run test (10MWRT). | baseline and up to month 24
  The 10MWRT is a timed functional test used to measure walking or running speed over 10 meters by the study population
Blood sorbitol levels | Baseline and up to 3 months.
  Patients with SORD Deficiency develop extremely high sorbitol levels in cells and tissues, as aldose reductase converts glucose to sorbitol which then cannot be converted into fructose by SORD. Sorbitol is known to be toxic to many cell types.
  The measurement of change in sorbitol will provide evidence of the efficacy of the treatment (AT-007) used in the study.

SECONDARY OUTCOMES:
Charcot Marie Tooth Functional Outcome Measure (CMT-FOM) | Baseline and up to month 24
  The CMT-Fom is a performance-based measure that assesses the functional ability of patients with CMT. Total and subdomain scores as well as individual components of the CMT-FOM, each as it's own secondary endpoint will be evaluated to detect change over time.
Charcot Marie Tooth Health Index (CMTHI) | Baseline and up to month 24
  The CMTHI is a disease-specific patient reported outcome that assesses disease burden in the study population. This will be used to assess patient-detected disease burden over time.
Exit Interview | To be completed at month 24
  A blinded assessment of the study population's perspective on the impact of disease on their lives and the benefit or perceived harm during the study.
Muscle Magnetic Resonance Imaging (MRI) | Baseline and up to month 24 month
  Patients will undergo MRI of their legs to evaluate the fat deposition and the muscle size, both CMT-related parameters of disease progression.
Blood Sorbitol Levels and Correlation with Clinical Outcomes | Baseline and up to month 24
  Patients with SORD Deficiency develop extremely high sorbitol levels in cells and tissues, as aldose reductase converts glucose to sorbitol which then cannot be converted into fructose by SORD. Sorbitol is known to be toxic to many cell types. Longitudinal correlation of sorbitol levels with different clinical outcomes will provide support for the role sorbitol plays in the disease progression of CMT-SORD, and will demonstrate correlation of sorbitol level with clinical outcomes benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Shy, MD, Study Chair — University of Iowa
Locations (10):
- United States (7):
  - University of Colorado, Aurora, Colorado
  - University of Miami, Coral Gables, Florida
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hassman Research Institute, Berlin, New Jersey
  - University of Rochester, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Axon Clinical, s.r.o., Prague, Prague, Czechia
- Fondazione IRCCS Istituto Neurologico "Carlo Besta", Milan, Milano, Italy
- University College of London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No